CLINICAL TRIAL: NCT06257290
Title: The Role of Platelet TLRs in Platelet Activation During VTE
Acronym: ROT-PLAT-VTE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 22CH400; 2023-A00448-37 (Other: ANSM)
Record Dates: First submitted 2024-02-06; First posted 2024-02-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism; VTE; sequelae; immunothrombosis; platelets; inflammatory receptors
MeSH Terms: conditions — Venous Thromboembolism; Thromboinflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — quantification of TLR2/TLR4 receptor expression by flow cytometry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Venous ThromboEmbolic (VTE) patients: a diagnosis of Venous ThromboEmbolic (VTE) less than 72 hours old at inclusion, with a follow-up of 3 to 6 months
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — at Day 1 - date of patient inclusion at time of VTE diagnosis
Biological: blood sample — at 6 months (in the patient follow-up)

SUMMARY:
Venous thromboembolic disease (VTE) is a frequent and potentially serious pathology. Therapeutic management has improved considerably over the last few decades, enabling the application of codified management in line with the recently updated French management recommendations.

One of the main remaining difficulties concerns VTE sequelae, mainly post-thrombotic syndrome after deep vein thrombosis, and post-pulmonary embolism syndrome after pulmonary embolism. The mechanisms leading to the absence of complete repermeabilization of vessels affected by Venous thromboembolic disease (VTE) are still poorly understood.

The concept of immunothrombosis, closely associating immunity, inflammation and thrombosis, could (in part) explain the appearance of these sequelae. Platelets appear to play a key role in the onset of sequelae: Platelets are known to be involved both in the onset of a VTE episode and in the inflammatory response. This involvement is illustrated by the expression of inflammatory receptors such as TLR (toll-like receptor) 2 and TLR4.

Th aim to investigate the role of platelets in the occurrence of sequelae, mainly via their role in the inflammatory response, in Venous thromboembolic disease (VTE) patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Venous ThromboEmbolic (VTE) / Proximal Deep vein thrombosis (DVT) of the lower limb and/or pulmonary embolism ≤ 72heures
* Patients are 18 years of age or older at diagnosis.
* Patients received informed written consent
* Patients benefiting from social security coverage

Exclusion Criteria:

* Diagnosis of Venous ThromboEmbolic (VTE) more than 72 hours old
* Isolated sub-segmental pulmonary embolism
* Patients on antiplatelet agents
* Patients on non-steroidal anti-inflammatory drugs (NSAIDs)
* Life expectancy > 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Venous ThromboEmbolic (VTE) patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
expression of TLR2/ TRL4 | at day1 and at 6 months
  The characteristic membrane profile of the inflammatory role of platelets is quantified by TLR2/TLR4 receptors expression using flow cytometry.
  This profile will be compared between patients with VTE sequelae (objectified during follow-up, and defined in accordance with good practice recommendations) 20,21 and patients without VTE sequelae.
  o A patient with sequelae corresponds to patients who will present during follow-up with a post-thrombotic syndrome (defined by a Villalta score greater than or equal to 5) and/or a post-pulmonary post-pulmonary embolism syndrome (defined by NYHA stage II, III or IV dyspnea, and the presence of perfusion perfusion sequelae on lung scintigraphy).

SECONDARY OUTCOMES:
Analysis of characteristic soluble profile of the inflammatory role of platelets | at day1 and at 6 months
  The characteristic soluble profile of the inflammatory role of platelets associated with the existence of sequelae remote from the acute episode of VTE, is quantified by blood assay of platelet immunomodulatory factors (ELISA technique): soluble CD62P, HMGB1, RANTES, PF4, soluble CD40L

CONTACTS AND LOCATIONS:
Locations (1):
- Chu St-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No